CLINICAL TRIAL: NCT04388891
Title: Clinical Feasibility of Minimally Supervised Therapy After Stroke With a Hand Rehabilitation Robot (ReHapticKnob): Pilot and Main Study
Brief Title: Clinical Feasibility of Minimally Supervised Therapy After Stroke With a Hand Rehabilitation Robot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Clinica Hildebrand Brissago (Other); Rehabilitation Engineering Laboratory, ETHZ (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ReHapticKnob 2020
Record Dates: First submitted 2020-05-05; First posted 2020-05-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Stroke; Hand impairment; Robot-assisted therapy; Minimally supervised therapy; Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally supervised therapy (Experimental): This group will undergo minimally supervised therapy with the robot ReHapticKnob.
  Interventions: Device: Minimally supervised therapy with the ReHapticKnob

INTERVENTIONS:
Device: Minimally supervised therapy with the ReHapticKnob — The therapy with the ReHapticKnob is performed in the clinic in addition to the conventional therapy. During the supervised and semi-supervised phases (first 2 weeks), the intervention dose is 5 sessions of approximately 45 minutes per week. During each session, the robot proposes a set of 3 exercises, each lasting between 10 and 15 minutes. During the minimally supervised phase (third and fourth week), the duration of the ReHapticKnob therapy is not specified, since the patient can decide by him/herself when to use the device, e.g. during freetime or during the weekend.

SUMMARY:
The ReHapticKnob is a robot for hand rehabilitation after stroke. We aim to investigate the feasibility of minimally supervised therapy with the ReHapticKnob with stroke patients in a rehabilitation clinic, evaluate the usability of the ReHapticKnob (user interface and implemented exercises which were adapted for independent usage), and quantify the dose of additional robotic therapy that patients perform in a minimally supervised setting.

Minimally supervised therapy means that after a training phase, where the therapists teach to the patients how to perform the exercises with the robot, the patients can autonomously train with the robot during free time without being directly supervised. Our hypothesis is that minimally supervised therapy might be a possible way to increase therapy dose for stroke patients, with the potential to further improve recovery of hand function with minimal additional burden for therapists and for the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Male and female stroke patients between 18 and 90 years old;
* pre-stroke Modified Rankin Score ≤ 1;
* acute/subacute stroke (within (≤) 6 weeks from onset);
* NIHSS ≥ 1 in at least one of the items regarding motor function, sensory functions and ataxia;
* the patient read, understood and signed the informed consent.

Exclusion Criteria:

* Modified Ashworth Scale > 2 for one or more of the following muscles: shoulder adductors, forearm pronator and supinator, flexors and extensors of elbow, wrist and fingers;
* moderate to severe aphasia: Goodglass-Kaplan scale < 3;
* moderate to severe cognitive deficits: levels of cognitive functioning-revised (LCF-R) < 8;
* functional impairment of the upper limb due to other pathologies;
* severe pain in the affected arm: visual analogue scale for pain (VASp) ≥ 5;
* other pathologies which may interfere with the study;
* pacemakers and other active implants.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Compliance as assessed by dose | Compliance to minimally supervised therapy is calculated at the end of the fourth week of the study protocol.
  Sum of the dose of robot-assisted therapy without direct supervision that the patient performs.

SECONDARY OUTCOMES:
Usability as assessed by the Post-Study System Usability Questionnaire | Usability is first measured at the end of the second week.
  Usability of the ReHapticKnob measured with the Post-Study System Usability Questionnaire (version 3). This questionnaire consists of 16 questions and the possible response options vary between 1 (strongly agree) and 7 (strongly disagree).
Usability as assessed by the Post-Study System Usability Questionnaire | Usability is measured again at the end of the fourth week.
  Usability of the ReHapticKnob measured with the Post-Study System Usability Questionnaire (version 3). This questionnaire consists of 16 questions and the possible response options vary between 1 (strongly agree) and 7 (strongly disagree).
Usability as assessed by the System Usability Scale | Usability is first measured at the end of the second week.
  Usability of the ReHapticKnob measured with the System Usability Scale. The possible response options vary between 1 (strongly disagree) and 5 (strongly agree).
Usability as assessed by the System Usability Scale | Usability is measured again at the end of the fourth week.
  Usability of the ReHapticKnob measured with the System Usability Scale. The possible response options vary between 1 (strongly disagree) and 5 (strongly agree).
Usability as assessed by the NASA Task Load Index | Usability is first measured at the end of the second week.
  Usability of the ReHapticKnob measured with the NASA Task Load Index.
Usability as assessed by the NASA Task Load Index | Usability is measured again at the end of the fourth week.
  Usability of the ReHapticKnob measured with the NASA Task Load Index.
Evolution of patient's satisfaction with robot-assisted therapy as assessed by a 5-point scale | First to fourth week.
  A 5-point scale is presented by the robot at the end of each therapy session to measure patient's satisfaction with robot-assisted therapy.
Change in upper limb functions as assessed by the Fugl-Meyer Assessment of Upper Extremities (FMA-UE) | Baseline functions are assessed at the beginning of the first week, final functions are assessed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) upper limb functions as assessed by the FMA-UE.
Change in upper limb functions as assessed by the ABILHAND | Baseline functions are assessed at the beginning of the first week, final functions are assessed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) upper limb functions as assessed by the ABILHAND scale.
Change in upper limb functions as assessed by the Box and Block (BBT) test | Baseline functions are assessed at the beginning of the first week, final functions are assessed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) upper limb functions as assessed by the BBT test.
Change in upper limb functions as assessed by the Motor Evaluation Scale for Upper Extremities in Stroke Patients (MESUPES) | Baseline functions are assessed at the beginning of the first week, final functions are assessed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) upper limb functions as assessed by the MESUPES. The scores can vary between 0 and 58, and a higher score means a better outcome.
Change in upper limb functions as assessed by the modified Ashworth Scale (mAS) | Baseline functions are assessed at the beginning of the first week, final functions are assessed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) upper limb functions as assessed by the mAS.
Change in the active Range of Motion (aROM) for grasping as assessed by a custom robotic assessment | Baseline aROM is assessed at the beginning of the first week, final aROM is assessed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) aROM for grasping, i.e. for hand opening and closing. This is measured by the robot with a custom assessment.
Change in the active Range of Motion (aROM) for forearm rotation as assessed by a custom robotic assessment | Baseline aROM is assessed at the beginning of the first week, final aROM is assessed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) aROM for forearm pronation and supination. This is measured by the robot with a custom assessment.
Change in hand proprioception as assessed by a custom robotic assessment measuring the minimum difference in length that a patient can perceive | The baseline assessment is performed at the beginning of the first week, the final assessment is performed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) hand proprioception, defined as the minimum difference in length that a patient can perceive (i.e. just noticeable difference). This is measured by the robot with a custom assessment.
Change in haptic perception as assessed by a custom robotic assessment measuring the minimum difference in stiffness that a patient can perceive | The baseline assessment is performed at the beginning of the first week, the final assessment is performed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) haptic perception, defined as the minimum difference in stiffness that a patient can perceive. This is measured by the robot with a custom assessment.
Monitoring of muscle tone | First to fourth week.
  Muscle tone will be monitored throughout the robot-assisted therapy with assessments embedded in some of the exercises implemented in the ReHapticKnob.
Change in knowledge about stroke and health as assessed by a custom questionnaire consisting of 20 open or multiple-choice questions about stroke and health | The baseline assessment is performed at the beginning of the first week, the final assessment is performed at the end of the fourth week.
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) knowledge about stroke and health, defined as the number of correct answers out of total number of questions asked about stroke and health. The questionnaire with the 20 questions about stroke and health is custom made.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Rossi, Dr. med., Principal Investigator — Clinica Hildebrand Brissago
Locations (1):
- Clinica Hildebrand Centro di riabiliazione Brissago, Brissago, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devittori G, Dinacci D, Romiti D, Califfi A, Petrillo C, Rossi P, Ranzani R, Gassert R, Lambercy O. Unsupervised robot-assisted rehabilitation after stroke: feasibility, effect on therapy dose, and user experience. J Neuroeng Rehabil. 2024 Apr 9;21(1):52. doi: 10.1186/s12984-024-01347-4. PMID 38594727
- [Derived] Devittori G, Ranzani R, Dinacci D, Romiti D, Califfi A, Petrillo C, Rossi P, Gassert R, Lambercy O. Progressive Transition From Supervised to Unsupervised Robot-Assisted Therapy After Stroke: Protocol for a Single-Group, Interventional Feasibility Study. JMIR Res Protoc. 2023 Nov 9;12:e48485. doi: 10.2196/48485. PMID 37943580